CLINICAL TRIAL: NCT01690728
Title: Effect of Physical Activity on Weight Loss and Cardiovascular Risk Factors After Gastric Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Responsible Party: Principal Investigator, Lene Hymøller Mundbjerg, M.D. PhD-student, Esbjerg Hospital - University Hospital of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CBR-001
Record Dates: First submitted 2012-09-14; First posted 2012-09-24 (Estimated); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Morbid Obesity; Inactivity
Keywords: Obesity; Gastric bypass
MeSH Terms: conditions — Obesity, Morbid; Sedentary Behavior; Obesity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physical Activity (Active Comparator): 40 min exercise supervised by physiotherapists two times weekly in six month.
  Interventions: Behavioral: Physical Activity
- Control Group (No Intervention): These participants follows the standard post surgery follow-up consisting of counseling by dietitians, nurses and doctors.

INTERVENTIONS:
Behavioral: Physical Activity — The intervention program will continue for six month consisting of two weekly sessions of 40 min exercise supervised by physiotherapists. The supervised exercise program will take place at the training center Fitness.dk in Esbjerg and Kolding. It will be in cooperation with physiotherapists at the Therapy Department of Sydvestjysk Sygehus Esbjerg and the Therapy Department of Fredericia and Kolding Sygehus, Sygehus Lillebælt. The exercise program at the two centers will be equal. In addition the patients will be provided with free access to a fitness center. The patient will be encouraged to do at least 3.5 hours of moderate to vigorous physical activity per week.
  Arms: Physical Activity

SUMMARY:
The aim of this study is to increase our knowledge about the effect of physical activity in patients who have undergone gastric bypass surgery. The study will provide novel information in two areas. The main objective is to study the effect of physical activity on the weight loss and cardiovascular risk factors. This will be accomplished in a randomized clinical trial in patients, who are eligible for gastric bypass (GB). Patients will be randomized to six month of structured physical activity or standard postoperative counseling. The study will include an exhaustive panel of blood tests related to cardiovascular risk and the most extensive evaluation of structural and functional vascular test done in this patient group so far. In addition the study will provide information of the effect of bariatric surgery per se since both pre- and postoperative investigations are conducted. The study will learn us to what degree it is possible to motivate this group of patients to increased physical activity. All together this will enable us to improve the counseling of the patients undergoing GB.

DETAILED DESCRIPTION:
The study will be conducted as a prospective, randomized, controlled, two-group, intervention study. Patients will be recruited among individuals referred to the tertiary center for bariatric surgery. The patients will be asked to participate in the study when they attend the preoperative education for bariatric surgery. Randomization will be performed in blocks ensuring an equal distribution of type 2 diabetes patients in the two study groups.

Participants will be investigated before gastric bypass surgery, six, 12 and 24 month post-operative. Intervention, consisting of structured physical activity will take place from six to 12 month after operation.

The intervention program will continue for six month. The supervised exercise program will take place at the training center consisting of 40 min. sessions two times pr. week for 26 consecutive weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 25 - 60 years
* Able to understand and cooperate with the interventions in the study
* Eligible for gastric bypass surgery

Exclusion Criteria:

* Inability to perform physical activity at the intensity and quantity required in the study, such as physical disabled patients including severe osteoarthritis
* Use of vitamin K antagonists, oral contraceptives, or hormone replacement therapy

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Weight loss | Measures 1-2 weeks before gastric bypass, change from baseline 6, 12 and 24 month post-surgery
  The participants pre-operative weight are measured before gastric bypass surgery. This measure will take place within 2 weeks before surgery. Weight change from baseline will be measured 6, 12 and 24 months post-surgery.

SECONDARY OUTCOMES:
Blood tests | Measures 1-2 weeks before gastric bypass, 6, 12 and 24 month post-surgery
  Exhaustive panel of blood tests related to cardiovascular risk. The participants are measured before gastric bypass surgery. This measure will take place within 2 weeks before surgery. Changes in blood analyses from baseline will be measured 6, 12 and 24 months post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Claus B Juhl, MD, ph.d., Principal Investigator — Esbjerg Hospital - University Hospital of Southern Denmark
Locations (1):
- Center of Bariatric Research, Dep. of Endocrinology, Hospital of South West Denmark, Esbjerg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stolberg CR, Mundbjerg LH, Bladbjerg EM, Funch-Jensen P, Gram B, Juhl CB. Physical training following gastric bypass: effects on physical activity and quality of life-a randomized controlled trial. Qual Life Res. 2018 Dec;27(12):3113-3122. doi: 10.1007/s11136-018-1938-9. Epub 2018 Jul 25. PMID 30046976
- [Derived] Stolberg CR, Mundbjerg LH, Funch-Jensen P, Gram B, Bladbjerg EM, Juhl CB. Effects of gastric bypass surgery followed by supervised physical training on inflammation and endothelial function: A randomized controlled trial. Atherosclerosis. 2018 Jun;273:37-44. doi: 10.1016/j.atherosclerosis.2018.04.002. Epub 2018 Apr 6. PMID 29677629
- [Derived] Mundbjerg LH, Stolberg CR, Cecere S, Bladbjerg EM, Funch-Jensen P, Gram B, Juhl CB. Supervised Physical Training Improves Weight Loss After Roux-en-Y Gastric Bypass Surgery: A Randomized Controlled Trial. Obesity (Silver Spring). 2018 May;26(5):828-837. doi: 10.1002/oby.22143. Epub 2018 Mar 22. PMID 29566463